CLINICAL TRIAL: NCT05584176
Title: Over the Counter Rapid Antigen Test for Detection of SARS-CoV-2 Virus: Clinical Evaluation
Brief Title: COVID-19 MP Biomedicals SARS-CoV-2 Ag OTC: Clinical Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MP Biomedicals, LLC (Industry)
Collaborators: New Day Diagnostics (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EDP-SOP-TNC-014
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Results first posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2022-10

CONDITIONS: SARS-CoV2 Infection; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is an open-label, prospective study to evaluate the sensitivity and specificity of the Rapid SARS-CoV-2 Antigen Test when a lay person conducts the test on themselves or another study participant. Potential subjects will be those presenting for COVID-19 testing. The study will evaluate the performance of the Rapid SARS-CoV-2 Antigen Test by comparing it to a high sensitivity EUA SARS-CoV-2 RT-PCR assay to calculate both the positive percent agreement (PPA, or sensitivity) and the negative percent agreement (NPA, or specificity).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Subject 14-65+ years of age (Experimental): Participants will have a nasopharyngeal swab sample collected by trained study site personnel for testing on a high sensitivity EUA SARS-CoV-2 RT-PCR assay to compare the result to the result of the Rapid SARS-CoV-2 Antigen Test. The participant will then self-collect or, if both are over 18, collect from another study participant an anterior nasal swab sample and test using the Rapid SARS-CoV-2 Antigen Test.
  Interventions: Device: iCura COVID-19 Antigen Rapid Home Test; Device: RT-PCR Test
- At least 30 children between 2 and 13 years of age (Experimental): Participants 2-13 years of age will have a nasopharyngeal swab sample collected by trained study site personnel for testing on a high sensitivity EUA SARS-CoV-2 RT-PCR assay to compare the result to the result of the Rapid SARS-CoV-2 Antigen Test. The parent or legal guardian of the child will collect an anterior nasal swab sample from the child and perform the Rapid SARS-CoV-2 Antigen Test.
  Interventions: Device: iCura COVID-19 Antigen Rapid Home Test; Device: RT-PCR Test

INTERVENTIONS:
Device: iCura COVID-19 Antigen Rapid Home Test — Candidate Ag self-test kit anterior nasal specimen collection and testing will be done under the supervision of qualified site personnel in person. Comparator NP samples shall be collected at least 15 minutes prior to Ag samples with at least 15 minutes between nasal collections including collections that may occur prior to study enrollment. Comparator samples will be collected first by qualified personnel at a study site or physician's office using an FDA authorized nasopharyngeal swab collection kit and SARS-CoV-2 molecular assay.
Device: RT-PCR Test — High sensitivity RT-PCR COVID-19 Test

SUMMARY:
SARS-CoV-2 rapid antigen over the counter clinical performance evaluation

DETAILED DESCRIPTION:
Coronavirus disease (COVID-19) is a disease caused by a newly discovered coronavirus, severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). The SARS-CoV-2 is a β-coronavirus, which is enveloped non-segmented positive-sense RNA virus 2. It is spread by human-to-human transmission via droplets or direct contact, and infection has been estimated to have mean incubation period of 6.4 days and a basic reproduction number of 2.24-3.58. Among patients with pneumonia caused by SARS-CoV-2, fever was the most common symptom, followed by cough. On 11 March 2020, the COVID-19 outbreak was characterized as a pandemic by the WHO. Since then, over 70 million people worldwide have been infected with the virus with over 1.5 million deaths attributed to the virus. Laboratory testing for SARS-CoV-2 is currently being performed to determine if an individual has active infection via detection of viral RNA or if an individual has an immune response to the virus from a previous infection via detection of antibodies.

Specimen collection is a crucial first step in the evaluation of an individual's SARS-CoV-2 infection status. The goal of this project is to evaluate a rapid SARS-CoV-2 antigen test for over the counter (OTC) use. Study subjects under EDP supervision, either in-person or via video conference, will collect and test anterior nasal swab samples and a Study Representative will collect and ship a second nasopharyngeal swab sample for comparator PCR testing. The Rapid SARS-CoV-2 Antigen Test collection and testing methodology is viewed as a convenient and inexpensive method to test clinical specimens for SARS-CoV-2 and OTC access will improve the availability of COVD-19 testing.

The COVID-19 Antigen Rapid Test Device detects SARS-CoV-2 viral antigens through visual interpretation of color development. Anti-SARS-CoV-2 antibodies are immobilized on the test region of the nitrocellulose membrane. Anti-SARS-CoV-2 antibodies conjugated to colored particles are immobilized on the conjugated pad. A sample is added to the extraction buffer which is optimized to release the SARS-CoV-2 antigens from specimen. During testing, the extracted antigens bind to anti-SARS-CoV-2 antibodies conjugated to colored particles. As the specimen migrates along the strip by capillary action and interacts with reagents on the membrane, the complex will be captured by the anti-SARS-CoV-2 antibodies at the test region. Excess colored particles are captured at the internal control zone. The presence of a colored band in the test region indicates a positive result for the SARS-CoV-2 viral antigens, while its absence indicates a negative result. A colored band at the control region serves as a procedural control, indicating that the proper volume of specimen has been added and membrane wicking is working.

ELIGIBILITY:
Inclusion Criteria:

* The study population will include subjects from 2 years old to greater than 65 years old.
* Lay subjects who perform the test on themselves must be able to read, write, speak, and understand English.

Exclusion Criteria:

* Subjects less than 2 years old will be excluded.
* Participants who regularly use home diagnostic tests, such as glucose meters, or are trained medical or laboratory professionals will be excluded.
* Persons under 14 years of age will be excluded from performing the Rapid SARS-CoV-2 Antigen Test on themselves.
* Persons under 2 years of age will be excluded from participation.
* Persons under 18 years of age will be excluded from performing the Rapid SARS-CoV-2 Antigen Test on another qualified participant.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Liggett, PhD., Principal Investigator — New Day Diagnostics
Locations (4):
- United States (4):
  - Accel Research, DeLand, Florida
  - Daniel Sarkis, Gainesville, Florida
  - Accel Research Site St. Petersburg, St. Petersburg, Florida
  - EDP Biotech Corporation, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rothan HA, Byrareddy SN. The epidemiology and pathogenesis of coronavirus disease (COVID-19) outbreak. J Autoimmun. 2020 May;109:102433. doi: 10.1016/j.jaut.2020.102433. Epub 2020 Feb 26. PMID 32113704
- [Background] Guo YR, Cao QD, Hong ZS, Tan YY, Chen SD, Jin HJ, Tan KS, Wang DY, Yan Y. The origin, transmission and clinical therapies on coronavirus disease 2019 (COVID-19) outbreak - an update on the status. Mil Med Res. 2020 Mar 13;7(1):11. doi: 10.1186/s40779-020-00240-0. PMID 32169119
- [Background] Lai CC, Shih TP, Ko WC, Tang HJ, Hsueh PR. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and coronavirus disease-2019 (COVID-19): The epidemic and the challenges. Int J Antimicrob Agents. 2020 Mar;55(3):105924. doi: 10.1016/j.ijantimicag.2020.105924. Epub 2020 Feb 17. PMID 32081636
- See also: Johns Hopkins University Center for Health Security Website. 2020. — https://www.centerforhealthsecurity.org
- See also: WHO. 2022. — https://www.who.int/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Subject 14-65+ Years of Age | At Least 30 Children Between 2 and 13 Years of Age
Started | 298 | 34
Completed | 298 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subject 14-65+ Years of Age | At Least 30 Children Between 2 and 13 Years of Age | Total
Number analyzed (Participants) | 298 | 34 | 332
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 34 | 34
  Between 18 and 65 years | 260 | 0 | 260
  >=65 years | 38 | 0 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 27 | 205
  Male | 120 | 7 | 127
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 13 | 41
  White | 196 | 15 | 211
  More than one race | 65 | 5 | 70
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 298 | 34 | 332

OUTCOME MEASURES:

1. Primary Outcome: Positive Percent Agreement
Description: The acceptance criteria for this study is Positive Percent Agreement (PPA) greater than or equal to eighty percent in a comparison between the Rapid SARS-CoV-2 Antigen Test and RT-PCR comparator test results. The PPA was defined as the proportion of true positive tests, defined by a concordant candidate and comparator test result of positive, out of all positive candidate test results.
Time Frame: One hour
Population: Of the 332 samples collected across four sites in Tennessee and Florida, 188 met inclusion/exclusion criteria and had valid comparator RT-PCR data including ct values from NP swabs. There were an additional 59 samples which met inclusion/exclusion criteria and have valid comparator RT-PCR data, but the comparator swabs were collected by AN swab instead of NP swab.
Measure: Count of Participants; unit: Participants
Arm/Group | Subject 14-65+ Years of Age | At Least 30 Children Between 2 and 13 Years of Age
Number analyzed (Participants) | 176 | 12
Participants | 53 | 2

2. Primary Outcome: Negative Percent Agreement
Description: The acceptance criteria for this study is Negative Percent Agreement (NPA) greater than or equal to ninety-eight percent in a comparison between the Rapid SARS-CoV-2 Antigen Test and RT-PCR comparator test results. The NPA was defined as the proportion of true negative tests, defined by a concordant candidate and comparator test result of negative, out of all negative candidate test results.
Time Frame: One hour
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Subject 14-65+ Years of Age | At Least 30 Children Between 2 and 13 Years of Age
Number analyzed (Participants) | 176 | 12
Participants | 123 | 10

3. Secondary Outcome: Detection of Asymptomatic Positives
Description: Number of participants with a positive PCR comparator result, but reported no symptoms or epidemiological reasons to suspect COVID-19 infection within the past 14 days. This will be compared to their Rapid SARS-CoV-2 Antigen Test result to determine the ability of the Rapid SARS-CoV-2 Antigen Test to detect individuals who are infected but are not symptomatic.
Time Frame: One hour
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Subject 14-65+ Years of Age | At Least 30 Children Between 2 and 13 Years of Age
Number analyzed (Participants) | 176 | 12
Participants | 3 | 0

ADVERSE EVENTS:
Time Frame: One hour
Description: This study was deemed to have a less than significant risk by IRB assessment, and not sites reported any adverse events during or after the study enrollment period.
Arm/Group | Subject 14-65+ Years of Age | At Least 30 Children Between 2 and 13 Years of Age
All-Cause Mortality (participants affected / at risk) | 0/298 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/298 | 0/34
Other Adverse Events (participants affected / at risk) | 0/298 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT05584176/Prot_003.pdf
  • Statistical Analysis Plan (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT05584176/SAP_005.pdf
  • Informed Consent Form: Informed Consent Form for Adults and Minors 14-17 Years (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/76/NCT05584176/ICF_001.pdf
  • Informed Consent Form: Informed Assent Form for Subjects 7-13 Years of Age (2021-11-04): https://cdn.clinicaltrials.gov/large-docs/76/NCT05584176/ICF_002.pdf